CLINICAL TRIAL: NCT02682147
Title: Functional CT Assessment of Pulmonary Arterial Dysfunction in Smoking Associated Emphysema
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eric A. Hoffman (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Eric A. Hoffman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201508782; R01HL130883 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-02-15 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sildenafil (Experimental): 40 subjects (20M and 20F) will be recruited to study non-contrast imaging at TLC and 20%VC and with contrast using DECT scans to assess perfused blood volume. For the intervention, the subject will be administered 20 mg of sildenafil and then the same scanning will be repeated one hour after sildenafil administration.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — One dose of 20 mg Sildenafil will be given one hour before CT imaging.
  Other Names: Revatio

SUMMARY:
This study will use dual energy x-ray computed tomography (DECT) to evaluate the relationship between heterogeneous perfusion, hypoxia (low oxygen in inspired gas) and induction of pulmonary vascular dilatation to characterize emphysema susceptibility in a normal smoking population. The investigators will correlate DECT measures of perfusion with lung injury measured by single photon emission computed tomography (SPECT). The investigators will study the effect of pulmonary arterial vasodilation to see if it eliminates indices of persistent lung injury in smokers that are susceptible to emphysema

DETAILED DESCRIPTION:
Imaging-based metrics have recently played a central role in the quest to identify chronic obstructive pulmonary disease (COPD) phenotypes, serving to establish homogeneous sub-populations to aid in genotyping, therapeutic targeting and design and outcomes assessment. Recent findings in both animals and humans have lead us to believe that CT derived perfusion (PBF) and mean transit time (MTT) measures within regionally injured lung parenchyma provide for a functional phenotype of which may be directly tied to the etiology of the pathologic process leading to emphysema in acentrilobular emphysema susceptible subset of the smoking population. The primary hypotheses of the proposal are built around the notion that smokers prone to emphysema have abnormal vasoregulation in that regional hypoxic pulmonary vasoconstriction (HPV) continues despite regional lung injury. This failure to block vasoconstriction alters the repair response and leads to tissue destruction in emphysema susceptible smokers (SS) with abnormal vasoregulation. The normal response to regional hypoxia is to shunt blood towards better-ventilated regions. However, smoking induces small scale, regional infiltrates which in turn lead to local hypoxia, HPV would interfere with defense mechanisms serving to clear the irritant and thus interfere with mechanisms of repair. The investigators have demonstrated that, in SS subjects with normal PFTs but CT evidence of early centriacinar emphysema (CAE), there is an increased heterogeneity of perfusion. This is supportive of the notion that attenuation of vasoconstriction has failed. Further, the investigators have demonstrated a tight correlation between quantitative CT evidence of emphysema with reduced lung volume (LV) filling down to very small amounts of emphysema.

The investigators outline a series of experiments seeking to:

1. link increased pulmonary perfusion heterogeneity in SS subjects to the lung's response to alveolar oxygenation;
2. establish that the perfusion heterogeneity is reversible;
3. demonstrate that the response to inflammation and not just inflammation itself is a key factor in the increased heterogeneity.

With any combination of positive outcomes of this study, the investigators will have provided new insights into disease etiology, serving to provide new targets for disease intervention and providing the tools needed for assessing outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 25 and 65.
2. Must be currently smoking at least 1/2 pack/day (confirmed with cotinine level).
3. Must have pulmonary function test (PFT) results that meet the following (there will be two groups):

   Group 1:
   * Forced expiratory volume at one second (FEV1)/Forced vital capacity (FVC) > 70%
   * Forced Expiratory Flow at 25-75% of predicted(FEF25-75) > 79% of predicted
   * FVC greater than 80% of predicted

   Group 2:

   For subjects with mild lung impairment:
   * FEV1>80% of predicted
   * FEV1/FVC<0.7
4. Must be able to give informed consent for self.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Body Mass Index (BMI) greater than 32.
3. Weight of greater than 220 pounds (100 kg).
4. Allergies to shell fish, seafood, eggs or iodine.
5. Heart disease, kidney disease or diabetes.
6. Diagnosis of asthma.
7. Usage of any medications that are known to affect the heart or lungs (contraceptives, anti-depressants, analgesics EXCEPT aspirin, antihypertensives, and medications for osteoporosis and gastrointestinal diseases will be allowed).
8. Any metal in or on the body between the nose and the abdomen.
9. Any major organ system disease (by judgment of study medical team).
10. A glomerular filtration rate of 60 cc per minute or less.

For the subjects that will receive Sildenafil as part of the study, additional exclusion criteria are as follows:

1. Nitroglycerin usage or nitrates (in addition to nitroglycerin) and use of phosphodiesterase 5 (PDE5) inhibitors within the previous 7 days of the study date.
2. Prior history of hypersensitivity to Sildenafil.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Perfused blood volume assessed pre and post sildenafil administration in susceptible smoker (SS) subjects. | Pre sildenafil adminstration and one hour after sildenafil adminstration.
  Regional heterogeneity perfused blood volume will be measured by duel energy CT scan at two time points and compared at two points, pre and post the administration of sildenafil.
Perfused blood volume assessed pre and post sildenafil administration in non-susceptible smoker (SS) subjects. | Pre sildenafil adminstration and one hour after sildenafil adminstration.
  Regional heterogeneity perfused blood volume will be measured by duel energy CT scan at two time points and compared at two points, pre and post the administration of sildenafil.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Hoffman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
CT images will be shared including non-contrast images at TLC, FRC and RV as well as dual energy CT image data used to assess regional perfused blood volume. All associated pulmonary function test results will be shared. CT-derived metrics
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available starting 6 months after publication of the primary results of each aim.
Access Criteria: Data will be provided to academic-based researchers upon written request to the PI, Eric A. Hoffman, PhD. A nominal charge will be made for the time it takes for a technician to prepare and transfer the requested data. This costs will not exceed $250. This service will be available for a minimum of 2 years of study close.

REFERENCES:
- [Result] Alford SK, van Beek EJ, McLennan G, Hoffman EA. Heterogeneity of pulmonary perfusion as a mechanistic image-based phenotype in emphysema susceptible smokers. Proc Natl Acad Sci U S A. 2010 Apr 20;107(16):7485-90. doi: 10.1073/pnas.0913880107. Epub 2010 Apr 5. PMID 20368443
- [Result] Iyer KS, Newell JD Jr, Jin D, Fuld MK, Saha PK, Hansdottir S, Hoffman EA. Quantitative Dual-Energy Computed Tomography Supports a Vascular Etiology of Smoking-induced Inflammatory Lung Disease. Am J Respir Crit Care Med. 2016 Mar 15;193(6):652-61. doi: 10.1164/rccm.201506-1196OC. PMID 26569033
- Available data/document: Individual Participant Data Set: Data Distribution — http://www.i-clic.uihc.uiowa.edu/